CLINICAL TRIAL: NCT01046279
Title: Hypertension Monitoring in Glioma Patients Treated With Bevacizumab
Status: Terminated | Type: Observational
Why Stopped: Problems with enrollement of patients, less patients than expected
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-1700
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Glioma Patients
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Urine Samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glioma Patient receiving Bevacizumab: Patients with histological diagnosis of anaplastic astrocytoma (WHO Grad III) or Glioma (WHO Grad IV)assigned to bevacizumab treatment (monotherapy or adjunctive to chemotherapy) for therapeutic reasons
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Patients with histological diagnosis of anaplastic astrocytoma (WHO Grad III) or Glioma (WHO Grad IV) assigned to bevacizumab treatment (monotherapy or adjunctive to chemotherapy) for therapeutic reasons

SUMMARY:
Prospective casecontrol study in glioma patients undergoing treatment with bevacizumab (Avastin). At present there are no data on the correlation between occurrence of arterial hypertension and clinical outcome in patients with glioma or anaplastic astrocytoma. We will investigate whether glioma patients developing hypertension under bevacizumab treatment have a better outcome in terms of progression free survival, response rate and overall survival than equally treated patients remaining normotensive. Moreover, we will describe the dynamics of change in blood pressure after administration of bevacizumab in those patients developing hypertension.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: Patients aged 18 or older with histological diagnosis of anaplastic astrocytoma (WHO grade III) or glioma (WHO grade IV) Assigned to bevacizumab treatment (monotherapy or adjunctive to chemotherapy) for therapeutic reasons by an oncologist Patients should be on a stable or decreasing dose of steroids Willingness and ability to comply with the protocol Patient should present with a KPS of >=70 Signed informed consent

Exclusion criteria: Previous anti-angiogenic drugs other than bevacizumab Allergy or hypersensitivity against bevacizumab Contraindications to bevacizumab according to the Summary of Product of Characteristics Unwillingness to comply with regular assessments of response and performance of study-related procedures Any condition considered relevant for proper performance of the study or risk to the patients, at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioma patients receiving bevacizumab
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypertension | Hypertension under treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Zimmerli, MD, Principal Investigator — University Hospital Zurich, Internal Medicine
Locations (1):
- University Hospital Zurich, Internal Medicine, Zurich, Canton of Zurich, Switzerland